CLINICAL TRIAL: NCT03562182
Title: Effect of Steroid Administration on Maternal Blood Levels of hLPCAT1 mRNA
Acronym: LPCAT1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Maurice-Andre Recanati, Assistant Professor, Clinical Educator, Wayne State University
Other Study IDs: 041717MP2F
Record Dates: First submitted 2018-05-09; First posted 2018-06-19 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Fetal Lung Maturity; Respiratory Distress Syndrome in Premature Infant
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Weeks
Biospecimen Retention: Samples With DNA — LPCAT1 mRNA extracted from maternal plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women Receiving Antenatal Steroids: Group 2: Determine how (and if) serum hLPCAT1 mRNA changes with administration of a course of steroids by measuring its plasma levels before, 24hrs after the first dose and 24hrs after the second dose of bethamethasone as well as one and two week after the first dose. This is accomplished through a simple blood draw. We seek to understand the effects of the 2nd dose of steroids and determine if, once the hLPCAT1 expression begins, does it continue or does it turn off again after some time from steroid administration.
  Interventions: Other: blood draw
- Normal Pregnancy Controls: 1) Group 1: Determine the plasma levels of hLPCAT1 mRNA in pregnant women from 32- 36+6/7 weeks gestation. This is accomplished through a simple blood draw. More specifically, we seek to find out, at what moment in gestation, expression spontaneously begins.
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — Blood draw (2.5mL) to assess mRNA LPCAT1 levels

SUMMARY:
Neonatal respiratory distress syndrome affects babies who are born preterm and requires them to be placed on a ventilator in the Intensive Care Unit. Over 15 million babies were born premature and these numbers have been increasing. It is caused by lungs which are still too immature to produce adequate amounts of surfactant. This surfactant reduces the alveolar surface tension and maintains the alveoli from collapsing. Collapsed alveoli prevent gas exchange and greatly increase work of breathing. Surfactant is a biochemical complex made up mostly of phospholipids such as phosphatidylcholine and phosphatidylglycerol and these, in turn, appear to be synthesized by lysophosphatidylcholine acyltransferase 1 (LPCAT 1). The investigators have previously established that hLPCAT1 mRNA in maternal serum correlates with lamellar body count, a well established clinical marker of fetal lung maturity.

DETAILED DESCRIPTION:
OBJECTIVES/AIMS

1. Group 1: Determine the serum levels of hLPCAT1 mRNA in pregnant women from 32- 36+6/7 weeks gestation. More specifically, to determine at what moment in gestation, expression spontaneously begins.
2. Group 2: Determine how (and if) serum hLPCAT1 mRNA changes with administration of a course of steroids by measuring its levels before, 24hrs after the first dose and 24hrs after the second dose of bethamethasone as well as one and two week after the first dose. The investigators seek to understand the effects of the 2nd dose of steroids and determine if, once the hLPCAT1 expression begins, does it continue or does it turn off again after some time from steroid administration.
3. Correlate measures of neonatal outcomes (Apgars, cord gases, need for NICU admission, need for respiratory support, need for ventilator) with levels of hLPCAT1 in labor.

METHODOLOGY The first group will consist of patients with normal pregnancies who present for routine prenatal care between 32- 36 6/7 weeks. Once consented and enrolled in the study, participants will give a small (half a teaspoon) blood sample every other week until reaching 37 weeks.

In group 2, pregnant women who present for rule-out preterm labor will be offered participation in the study. Blood samples will be collected along with all other relevant clinical labs (in PAX gene tubes) on admission, 24hrs and 48hrs after the course of steroids is initiated. Samples will also be collected 1 and 2 weeks later to see if steroid effect degrades over time. This would have immense clinical implication, especially when it comes to rescue doses.

Investigators will also correlate measures of neonatal outcomes (such as apgar scores, blood gases, NICU admission, need to go on respiratory/ventilator support) to the most recent maternal serum hLPCAT1 throughout the study. If the patient delivers more than one week from the last sample, an hLPCAT1 will be acquired during labor.

Women with singleton pregnancies and no evidence of diabetes, hypertension, smoking, BMI > 35, Hgb < 10 g/dl or other confounding variables will be admitted to the study. In addition a baseline for hLPCAT1 maternal serum mRNA will be established by testing women from 32 - 36 +6/7 weeks gestation. All tests will consist of a half teaspoon (2.5 ml) blood collection using PAX gene tubes.

Consent will be obtained by the PI/Co-PI's and by residents/fellows and the signed consent sheet will become part of the chart. No remuneration will be offered. Investigators will seek 80 volunteers for this study, anticipating an approximate drop-out rate of 50% because of compliance issues and early deliveries.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy, no evidence of diabetes, hypertension, smoking, BMI > 35, Hgb < 10 g/dl or other confounding variables

Exclusion Criteria:

* Smoking, abnormal gestation, multiple gestatio

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Patients who seek obstetrical care at Wayne State/DMC
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Change in LPCAT1 mRNA levels in maternal plasma after antenatal steroid administration | The time points will be a baseline before steroids, 24h after the first dose, 24h after the second dose, a week after steroids and two weeks after steroids.
  The investigators will measure the level of LPCAT1 mRNA in maternal plasma before and after the administration of antenatal steroids.

SECONDARY OUTCOMES:
Number of participants admitted to the NICU with high LPCAT1 mRNA levels | Through study completion, within 2 months
  Maternal levels of LPCAT1 mRNA will be measured in labor and compared to the need for admission to NICU. Data gathered from a chart review.
Correlate the LPCAT1 mRNA copy number to need for intubation in the nicu | Through study completion, within 2 months
  LPCAT1 mRNA levels in labor will be correlated to need for intubation. Data gathered from a chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Recanati, MD, Principal Investigator — Assistant Professor OBGYN
Locations (1):
- Detroit Medical Ceter, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Result] Welch RA, Recanati MA, Welch KC, Shaw MK. Maternal plasma LPCAT 1 mRNA correlates with lamellar body count. J Perinat Med. 2018 May 24;46(4):429-431. doi: 10.1515/jpm-2017-0057. PMID 28926341
- [Result] Harayama T, Shindou H, Shimizu T. Biosynthesis of phosphatidylcholine by human lysophosphatidylcholine acyltransferase 1. J Lipid Res. 2009 Sep;50(9):1824-31. doi: 10.1194/jlr.M800500-JLR200. Epub 2009 Apr 21. PMID 19383981
- [Result] Welch RA, Shaw MK, Welch KC. Amniotic fluid LPCAT1 mRNA correlates with the lamellar body count. J Perinat Med. 2016 Jul 1;44(5):531-2. doi: 10.1515/jpm-2015-0008. PMID 25968427
- [Result] Ellis B, Kaercher L, Snavely C, Zhao Y, Zou C. Lipopolysaccharide triggers nuclear import of Lpcat1 to regulate inducible gene expression in lung epithelia. World J Biol Chem. 2012 Jul 26;3(7):159-66. doi: 10.4331/wjbc.v3.i7.159. PMID 22905292